CLINICAL TRIAL: NCT04002830
Title: A Multicenter, Safety and Efficacy Study of Taliglucerase Alfa in Subjects With Type 3 Gaucher Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ari Zimran (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Ari Zimran, PI, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI224302
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Gaucher Disease, Type 3
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Intervention Model Description: Type 3 Gaucher disease patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Taliglucerase Alpha (Experimental): Intravenous infusion of Taligluucerase alfa (Elelyso) in treatment-naive patients with type 3 Gaucher disease
  Interventions: Drug: Elelyso

INTERVENTIONS:
Drug: Elelyso — Taliglucerase alfa is currently an approved therapy in the United States and many other countries for adults and children with a confirmed diagnosis of Type 1 GD ,and is also approved for use in Type 3 GD in a small number of countries.
  Other Names: Taliglucerase Alfa

SUMMARY:
This is a multicenter study to assess the safety and efficacy of taliglucerase alfa (60 units/kg) in previously untreated subjects of any age with Type 3 GD. Subjects will receive an infusion of taliglucerase alfa every 2 weeks for 12 months. Subjects who tolerate the infusions well, and who are treated in centers where home therapy is the SOC will be allowed to switch from site to home treatment at the discretion of the PI but after no less than 3 uneventful infusions at the site.

DETAILED DESCRIPTION:
Patients with Type 3 GD exhibit both visceral and neurologic manifestations. In addition to the progressive neurologic involvement, somatic disease manifestations, especially splenomegaly and resulting cytopenia, contribute to significant mortality and morbidity . The effects of enzyme replacement therapy (ERT) on patients with Type 1 GD have been clearly documented and have a beneficial effect on visceral and hematologic disease parameters . It is known that recombinant enzyme does not pass the blood-brain barrier and has no effect on neurologic involvement . Probably due to the rarity of Type 3 GD, information on the somatic effects of ERT is largely limited to case reports or single-center series. There are also few reviews of cohorts but the clinical subtype, age, genotype, ERT dosage, accompanying therapies, and treatment response vary widely among patients in these cohorts. This prospective study aims to objectively evaluate the hematologic and visceral effects of ERT with taliglucerase alfa on a rather clinically and genetically homogenous group of treatment-naïve patients with Type 3 GD . For the purposes of this study, subjects receiving no Gaucher-specific medications for at least 12 months will be considered "untreated". The results of this study are expected to provide a more objective view of the degree of response of this patient type, and potentially create new areas of research.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any age; however, if female:

   * must be using contraception if of childbearing potential or must be surgically sterile
   * must not be lactating
2. Diagnosis of Type 3 GD by enzyme and sequence analysis; and confirmed by the Medical Monitor.
3. Splenomegaly at least 5 x multiples of normal (MN).
4. Treatment-naïve.

Exclusion Criteria:

Eligible subjects may not have any of the following exclusion criteria:

1. Type 2 GD.
2. Presence of myoclonic seizures.
3. At least one allele of:

   * N370S (N409S in recent nomenclature)
   * R496H (R535H in recent nomenclature)
4. Presence of calcification in heart valves or arteries in echocardiography.
5. Presence of untreated iron, folic acid, vitamin B12 deficiency and/or hypothyroidism. (Resolved anemia is not an exclusion criterion.)
6. Presence of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and/or hepatitis C infections.
7. Splenectomy and bone marrow transplantation.
8. Presence of any medical, emotional, behavioural, or psychological condition that in the judgment of the Investigator would interfere with the subject's compliance with the requirements of the study.
9. Any other disorder that may interfere with the results of the efficacy endpoints.
10. Pregnancy or breastfeeding.
11. Currently taking another investigational drug for any condition or any therapeutic drug for Gaucher disease.
12. The subject and/or subject's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the study.
13. Medical history of any food/drugs allergy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, Prof., Principal Investigator — Shaare Zedek Medical Center
Locations (3):
- All India Institute of Medical Sciences, New Delhi, India
- Shaare Zedek Medical Center, Jerusalem, Israel
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If a patient did not meet the inclusion criteria or meet any of the exclusion criteria listed in the protocol, the patient was excluded at screening visits and was not enrolled.
Groups:
- Taliglucerase Alfa: The intervention: Taliglucerase alfa (60 units/kg, intravenously, every 2 weeks for 12 months).
  The target population: Treatment-naïve subjects with Type 3 Gaucher Disease. Any subgroup considerations: All participants will receive the investigational product.
Period: Overall Study
Arm/Group | Taliglucerase Alfa
Started | 14 (All patients received 60U/kg every two weeks)
Completed (All patients received 60U/kg every two weeks) | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Taliglucerase Alfa: Intravenous infusion of Taligluucerase alfa (Elelyso) in treatment-naive patients with type 3 Gaucher disease
  Elelyso: Taliglucerase alfa is currently an approved therapy in the United States and many other countries for adults and children with a confirmed diagnosis of Type 1 GD ,and is also approved for use in Type 3 GD in a small number of countries.
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 3.2 [1.3 to 9.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 1
  India | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Spleen Volume Measured by MRI
Description: Percent change from baseline
Time Frame: from baseline to month 12
Measure: Median (Standard Error); unit: Percent change
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
Percent change | -51.33 (8.67)

2. Secondary Outcome: Percent Change From Baseline in Liver Volume Measured by MRI
Description: Percent change from baseline
Time Frame: from baseline to month 12
Measure: Median (Standard Error); unit: Percent change
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
Percent change | -33.91 (3.81)

3. Secondary Outcome: Percent Change in Hemoglobin
Description: Percent change from baseline
Time Frame: from baseline to Months 3, 6, 9, and 12
Measure: Median (Standard Error); unit: percentage change in hemoglobin (%)
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
percentage change in hemoglobin (%)
  3 months | 26.43 (7.92)
  6 months | 28.97 (6.43)
  9 months | 29.93 (6.50)
  12 months | 35.81 (8.88)

4. Secondary Outcome: Percent Change in Platelet Count
Description: Percent change from baseline
Time Frame: from baseline to Months 3, 6, 9, and 12
Measure: Median (Standard Error); unit: percentage change in platelet count (%)
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
percentage change in platelet count (%)
  3 months | 2.50 (66.09)
  6 months | 53.33 (56.20)
  9 months | 94.44 (54.20)
  12 months | 122.44 (79.82)

5. Secondary Outcome: Percent Change in Lyso-GB1
Description: Percent change from baseline
Time Frame: from baseline to Months 3, 6, 9, and 12
Measure: Median (Standard Error); unit: percentage change in Lyso-Gb1 (%)
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 14
percentage change in Lyso-Gb1 (%)
  3 months | -29.16 (3.99)
  6 months | -46.57 (7.95)
  9 months | -60.00 (4.16)
  12 months | -74.32 (5.60)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Taliglucerase Alfa
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa (N=14)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Upon recovery from general anesthesia for abdominal MRI per protocol, the patent developed shortness of breath, stridor and bleeding from the mouth, which lead to an overnight observation and treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa (N=14)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomitting (Gastrointestinal disorders) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Labored breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Suffocation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Mosquito bite (Injury, poisoning and procedural complications) | 1 (1)
Hypotonus (Nervous system disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pectus carinatum (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT04002830/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04002830/SAP_001.pdf